CLINICAL TRIAL: NCT00792038
Title: Effect of Cognitive Behavioral Therapy in OCD Highlighted by Neuropsychological Tests and MRI: Pathophysiology and Treatment Outcome Predictors
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: M-20080161
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Psychological tests; Magnetic Resonance Imaging; Cognitive therapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Full blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: OCD patients
- 2: Normal Controls

SUMMARY:
OCD patients are assessed before and after treatment using diagnostic tools, rating scales neuropsychological assessment and functional and structural MR-scans.

ELIGIBILITY:
Inclusion Criteria:

1. Steady state medication 3 months prior to the study

Exclusion Criteria:

1. History of head trauma or other organic brain disease
2. Pregnancy.
3. Pacemaker or other ferromagnetic materials in the body.
4. Comorbid psychiatric illnesses assessed using SCAN- interview (30) other than moderate depression (Ham-D<17) or anxiety disorders.
5. Antipsychotics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: OCD patients from the primary care clinics in middle Jutland, Denmark
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2009-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Y-Bocs | Before and after treatment approx 20 weeks apart

CONTACTS AND LOCATIONS:
Overall Officials: Tue BH Hartmann, Principal Investigator — Aarhus University Hospital, Risskov; Sanne Kjær, Study Director — Aarhus University Hospital, Risskov
Locations (1):
- Aarhus University Hospital, Risskov, Risskov, Denmark

REFERENCES:
- [Derived] Vandborg SK, Hartmann TB, Bennedsen BE, Pedersen AD, Thomsen PH. Memory and executive functions in patients with obsessive-compulsive disorder. Cogn Behav Neurol. 2014 Mar;27(1):8-16. doi: 10.1097/WNN.0000000000000021. PMID 24674961